CLINICAL TRIAL: NCT05630014
Title: Development and Piloting of a Family-Centered, mHealth-Enhanced Intervention to Promote Caregiving Mastery in Detection, Prevention, and Management of Delirium Superimposed on Dementia
Brief Title: Study of the Aliviado DSD Caregiving Mastery Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-01093
Record Dates: First submitted 2022-11-18; First posted 2022-11-29 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Delirium Superimposed on Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Family Caregivers of PLWD at High Risk for Delirium (Experimental): Participants will complete the Aliviado DSD Caregiving Mastery Program. This involves a caregiver education/training period from Week 0 to Week 2, and an implementation period from Week 3 to Week 6.
  Interventions: Behavioral: Aliviado DSD Caregiving Mastery Program

INTERVENTIONS:
Behavioral: Aliviado DSD Caregiving Mastery Program — Family caregiver intervention consisting of mHealth-app based educational videos and articles; caregiver-administered assessment tools and care plans; and motivational push notification reminders and encouragements.

SUMMARY:
Delirium superimposed on dementia (DSD) is an acute and serious condition that is common in persons living with dementia (PLWD). Involvement of family caregivers may aid prevention, early detection, and management of DSD. The purpose of the proposed study is two-fold. First, the investigators will develop a family-centered, mHealth-enhanced DSD caregiving mastery program ("Aliviado DSD Caregiving Mastery Program") through a 5-week co-design workshop with 8 family caregivers (Aim 1). The investigators will adapt/refine the existing clinician-centered DSD contents and an mHealth app from the evidence-based "Aliviado Dementia Care" program for use by family caregivers to support their day-to-day implementation of DSD detection, prevention, and management tasks in the community. Second, the investigators will pilot test the full Aliviado DSD Caregiving Mastery Program with family caregivers of PLWD at high risk for delirium, assessing feasibility, acceptability, app usability, and preliminary program impact (Aim 2).

ELIGIBILITY:
Inclusion Criteria:

To be eligible as a "dementia caregiver" in the co-design workshop, an individual must:

* be at least 18 years old,
* be English-speaking,
* provide at least 8 hours of unpaid care weekly or live with a community-dwelling PLWD,
* self-identify as unfamiliar with DSD,
* have the capacity to consent, and
* have Internet access

To be eligible as a "DSD caregiver" in the co-design workshop, an individual must:

* be at least 18 years old,
* be English-speaking,
* be a current or past dementia caregiver with experience caring for a relative or friend during his/her DSD episode within the past 12 months,
* have the capacity to consent, and
* have Internet access.

To be eligible to participate in the feasibility trial, an individual must meet all of the following criteria:

* Being 18 years old or older,
* English-speaking,
* Providing at least 8 hours of unpaid care per week to, or living with, a community dwelling PLWD whose Delirium Risk Assessment Score >=5,
* Having the capacity to give informed consent, and
* Having a smartphone with Internet access.

Exclusion Criteria:

* Individuals who are blind or deaf will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Yin Lin, Principal Investigator — NYU Rory Meyers College of Nursing
Locations (2):
- United States (2):
  - NYU Langone Health, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: [SL199@nyu.edu]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access to the data upon reasonable request. Requests should be directed toSL199@nyu.edu. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Focus Groups were conducted in Aim 1 with 8 family caregivers to develop the program. These participants were not considered enrolled for the purposes of this study.
Period: Overall Study
Arm/Group | Family Caregivers of PLWD at High Risk for Delirium
Started | 32
Completed | 26
Not Completed | 6
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: Of the 32 consented primary family caregivers, 2 did not meet the eligibility criteria and were excluded from all data analyses.
Arm/Group | Family Caregivers of PLWD at High Risk for Delirium
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: years] | 58.3 [34 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Complete the Study
Description: Measure of feasibility. Feasibility indicated by retention rate of 85%.
Time Frame: Week 6
Population: All eligible enrolled primary family caregivers (n = 30) were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Family Caregivers of PLWD at High Risk for Delirium
Number analyzed (Participants) | 30
Participants | 26

2. Primary Outcome: Program Satisfaction Questionnaire Score: Satisfaction
Description: Measure of acceptability. Acceptability was indicated by at least 80% of caregivers reporting high satisfaction. The questionnaire comprised 16 items, including 12 Likert-type questions assessing program satisfaction, one Yes/No question assessing caregivers' intention to make changes in how they provide care for PLWD based on what they learned from the program, and three open-ended questions for additional feedback. Each Likert-type item was rated on a 4-point scale (1 = strongly disagree; 2 = disagree; 3 = agree; 4 = strongly agree). The total satisfaction score was calculated as the sum of the 12 Likert-type items, yielding a possible range of 12-48, with higher scores indicating greater satisfaction (high satisfaction defined as a score > 36). This outcome is measured as the number of participants with a high satisfaction score.
Time Frame: Week 6
Population: All eligible primary caregivers who completed the study and the program satisfaction questionnaire (n = 26) were included in the analysis. One primary caregiver had a missing response on one Likert-type item; therefore, the total program satisfaction score was calculated as the average of the 11 completed Likert-type items multiplied by 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Family Caregivers of PLWD at High Risk for Delirium
Number analyzed (Participants) | 26
Participants | 26

3. Primary Outcome: Program Satisfaction Questionnaire Score: Intention to Change
Description: Measure of acceptability. Acceptability was indicated by at least 80% of caregivers responding "Yes" to the Yes/No question on the Program Satisfaction Questionnaire: "Will you make any changes in how you care for your relative or friend with dementia based on what you learned in this program?" This outcome is measured as the number of participants who answer "Yes" to the intention-to-change question.
Time Frame: Week 6
Population: All eligible primary caregivers who completed the study and the intention-to-change question on the program satisfaction questionnaire (n = 26) were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Family Caregivers of PLWD at High Risk for Delirium
Number analyzed (Participants) | 26
Participants | 26

4. Primary Outcome: Number of Participants Who Complete All Training Videos by Week 2
Description: Measure of acceptability.
Time Frame: Up to Week 2
Population: All eligible enrolled primary family caregivers (n = 30) were analyzed. One caregiver refused to complete the training videos and subsequently declined continued participation in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Family Caregivers of PLWD at High Risk for Delirium
Number analyzed (Participants) | 30
Participants | 29

5. Primary Outcome: Number of Participants Who Complete Weekly Delirium Screening at Least Twice by Week 6
Description: Measure of acceptability.
Time Frame: Up to Week 6
Population: All eligible enrolled primary family caregivers who completed the study (n = 26) were analyzed. Four eligible primary family caregivers dropped out of the study (n=3) or were lost to follow-up (n=1) before Week 6 and were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Family Caregivers of PLWD at High Risk for Delirium
Number analyzed (Participants) | 26
Participants | 26

6. Primary Outcome: Modified IBM Computer Usability Satisfaction Questionnaire Score
Description: Modified by the Aliviado team to assess the usability of mobile apps, it consists of (1) 22 Likert-type questions rated on a scale from 1 to 5 (1="Strongly Disagree"; 2 ="Disagree"; 3="Neither agree or disagree"; 4="Agree" 5="Strongly Agree") assessing app usability, content, and interface; (2) one 4-point item on readiness to launch; (3) three Yes/No questions assessing frequency of app use and internet connectivity; and (4) three open-ended questions to provide additional feedback. The total usability satisfaction score is calculated by averaging responses to the twenty-two 5-point Likert-type items related to app usability, content, and interface. A score of 4 or higher indicates high user satisfaction and good usability.
Time Frame: Up to Week 6
Population: Eligible primary caregivers who completed both the baseline and Week 6 assessments (n = 26) were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Family Caregivers of PLWD at High Risk for Delirium
Number analyzed (Participants) | 26
score on a scale | 4.41 [3.90 to 4.70]

7. Secondary Outcome: Change From Baseline in Caregiver Delirium Knowledge Questionnaire Score at Week 2
Description: 19-item assessment of caregivers' delirium knowledge. Item response options include "yes," "no," and "I don't know." Correct responses receive a score of 1, incorrect responses receive a score of 0. The total score ranges from 0-19; higher scores indicate greater delirium knowledge.
Time Frame: Baseline, Week 2
Population: Of the 33 enrolled caregivers, 29 eligible primary caregivers were included for analysis. Of the 4 excluded caregivers, 2 did not meet study eligibility, 1 was a secondary caregiver, and 1 primary caregiver withdrew before completing the Week 2 Caregiver Delirium Knowledge Questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Caregivers of PLWD at High Risk for Delirium
Number analyzed (Participants) | 29
score on a scale | 3.86 (3.61)

8. Secondary Outcome: Change From Baseline in Caregiver Delirium Knowledge Questionnaire Score at Week 6
Description: as for outcome 7
Time Frame: Baseline, Week 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Caregivers of PLWD at High Risk for Delirium
Number analyzed (Participants) | 26
score on a scale | 3.81 (3.57)

9. Secondary Outcome: Change From Baseline in Modified Caregiver Strain Index Score at Week 6
Description: 13-item assessment of strain related to care provision. Items are scored on a Likert scale from 0 (no) to 2 (Yes, on a regular basis). The total score is the sum of responses and ranges from 0 to 26; higher scores indicate greater strain.
Time Frame: Baseline, Week 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Caregivers of PLWD at High Risk for Delirium
Number analyzed (Participants) | 26
score on a scale | 0.04 (10.74)

10. Secondary Outcome: Change From Baseline in Center for Epidemiological Studies Depression Scale (CES-D) Score at Week 6
Description: 20-item assessment of symptoms of depression over the past 7 days. The total score ranges from 0 to 60, with higher scores indicating the presence of more symptomatology.
Time Frame: Baseline, Week 6
Population: Eligible primary caregivers who completed both the baseline and Week 6 assessments (n = 26) were included in the analysis. One caregiver had two missing values in the baseline assessment; therefore, the total baseline CES-D score for this caregiver was calculated as the average of the sum of the 18 answered items multiplied by 20.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Caregivers of PLWD at High Risk for Delirium
Number analyzed (Participants) | 26
score on a scale | -2.15 (6.66)

11. Secondary Outcome: Change From Baseline in Short Form Zarit Burden Interview Score at Week 6
Description: 12-item assessment of caregiver burden. Items are scored on a Likert scale from 0 (never) to 4 (nearly always). The total score is the sum of responses and ranges from 0 to 48. A score of 0-10 indicates no to mild burden; 10-20 indicates mild to moderate burden; and greater than 20 indicates high burden.
Time Frame: Baseline, Week 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Caregivers of PLWD at High Risk for Delirium
Number analyzed (Participants) | 26
score on a scale | -2.15 (4.82)

12. Secondary Outcome: Change From Baseline in DSD Caregiving Mastery Assessment Score (Competence) at Week 2
Description: 4-item DSD Competence Scale modified from Pearline's Competence Scale. Each item is rated on a scale from 1-4. The total score is the sum of responses and ranges from 4 to 16. Higher scores indicate greater levels of mastery.
Time Frame: Baseline, Week 2
Population: Eligible Primary caregivers who completed both the baseline and Week 2 assessments (n = 29) were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Caregivers of PLWD at High Risk for Delirium
Number analyzed (Participants) | 29
score on a scale | 1.62 (2.87)

13. Secondary Outcome: Change From Baseline in DSD Caregiving Mastery Assessment Score (Competence) at Week 6
Description: as for outcome 12
Time Frame: Baseline, Week 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Caregivers of PLWD at High Risk for Delirium
Number analyzed (Participants) | 26
score on a scale | 2.73 (3.38)

14. Secondary Outcome: Change From Baseline in DSD Caregiving Mastery Assessment Score (Self-Efficacy) at Week 2
Description: 25-item DSD self-efficacy scale developed by the Aliviado team to assess confidence of DSD prevention, detection, and management tasks. Each item is rated on a scale from 0-100. The total score is the average of sum of non-missing responses and ranges from 0 to 100. Higher scores indicate greater levels of mastery.
Time Frame: Baseline, Week 2
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Caregivers of PLWD at High Risk for Delirium
Number analyzed (Participants) | 29
score on a scale | 3.59 (10.1)

15. Secondary Outcome: Change From Baseline in DSD Caregiving Mastery Assessment Score (Self-Efficacy) at Week 6
Description: as for outcome 14
Time Frame: Baseline, Week 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Caregivers of PLWD at High Risk for Delirium
Number analyzed (Participants) | 26
score on a scale | 6.6 (10.17)

ADVERSE EVENTS:
Time Frame: Week 7 (Up to 30 Days Post-Study Completion).
Description: Systematic: All AEs and SAEs were based on caregiver reports in response to questions on standard AE and SAE forms.
  Non-systematic: Caregivers were encouraged to report any additional AEs and SAEs to the study team for up to 30 days post-completion.
Arm/Group | Family Caregivers of PLWD at High Risk for Delirium
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 1/26
Other Adverse Events (participants affected / at risk) | 4/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Family Caregivers of PLWD at High Risk for Delirium (N=26)
Emergency Room Visit (Musculoskeletal and connective tissue disorders) | 1 — The caregiver had an overnight ER visit because she tore a ligament in her hip while lifting.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Family Caregivers of PLWD at High Risk for Delirium (N=26)
Fever (Infections and infestations) | 1
Sinus infection (Infections and infestations) | 1
Increased physical symptoms (Infections and infestations) | 1 — Increased physical symptoms and feeling under the weather, likely cold symptoms.
Soreness and aches (Musculoskeletal and connective tissue disorders) | 1 — Arm soreness and hip and leg aches due to lifting the care recipient after a fall.
Migraines (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-28): https://cdn.clinicaltrials.gov/large-docs/14/NCT05630014/Prot_SAP_000.pdf